CLINICAL TRIAL: NCT00411216
Title: Recovery of Visual Acuity in Vestibular Deficits
Brief Title: Recovery of Visual Acuity in People With Vestibular Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Susan Herdman, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00000336; R01DC003196 (NIH)
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Vestibular Neuronitis; Vestibular Neuronitis, Bilateral; Vestibular Schwannoma
Keywords: vestibular rehabilitation; vestibular hypofunction
MeSH Terms: conditions — Vestibular Neuronitis; Neuroma, Acoustic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercises for gaze stabilization (Experimental): Experimental group performed vestibular adaptation and substitution exercises
  Interventions: Other: gaze stabilization exercises
- Control exercises (Placebo Comparator): Saccadic eye movements against a Ganzfeld to prevent retinal slip error signal; no head movements
  Interventions: Other: Control exercises

INTERVENTIONS:
Other: Control exercises — saccadic eye movements against a plain background; no head movements
  Arms: Control exercises
Other: gaze stabilization exercises — adaptation and substitutin exercises encorporating retinal lsip and head movements
  Arms: exercises for gaze stabilization

SUMMARY:
The purpose of this study is to determine whether exercises relieve the symptoms of dizziness and imbalance in people with vestibular deficits and improves the ability to see clearly during head movements. We hypothesize that the performance of specific adaptation and substitution exercises will result in an improvement in visual acuity during head movements while those patients performing placebo exercises will show no improvement.

DETAILED DESCRIPTION:
Decrements in visual acuity during head movement in patients with vestibular hypofunction are potentially serious problems. This deficit could contribute to decreased activity level, avoidance of driving with resultant diminished independence and, ultimately, limited social interactions and increased isolation. Oscillopsia occurs because of inadequate vestibulo-ocular reflex (VOR) gain and suggests that compensation for the vestibular loss has not occurred. The purpose of this study was to examine the effect of an exercise intervention on visual acuity during head movement in patients with unilateral and bilateral vestibular hypofunction. We hypothesized that 1) patients performing vestibular exercises would have improved visual acuity during head movement compared to patients performing placebo exercises; 2) there would be no correlation between dynamic visual acuity (DVA) and the patients' subjective complaints of oscillopsia; and 3) improvement in DVA would be reflected by changes in residual vestibular function as indicated by an increase in VOR gain.

Patients are assigned randomly to either the vestibular exercise or placebo exercise group. The randomization schedule is generated using a computer program for 2-sample randomization. The sequence was not concealed from the investigator who obtained consent from the subjects and supervised the exercises (SJH). The group assignment (vestibular exercise or placebo exercise) was concealed from the participants and from the investigator who performed the outcome measures.

The vestibular exercise group practiced exercises that consisted of adaptation exercises and eye-head exercises to targets (Table 1), which were designed to improve gaze stability 16. They also performed gait and balance exercises. The placebo exercise group performed exercises designed to be 'vestibular-neutral'.

ELIGIBILITY:
Inclusion Criteria:

* Patient had to have either a unilateral vestibular or bilateral vestibular hypofunction defined as follows: Unilateral vestibular deficits were defined by a > 25% difference in slow phase eye velocity between right and left sides on either the caloric or rotary chair test. Bilateral vestibular deficits were defined included refixation saccades made in response to unpredictable head thrusts to the right and left, a gain < .1 on rotary chair step test and a peak slow phase eye movement of <5 degrees/sec during irrigation of each ear on bithermal water caloric testing
* Healthy subjects with normal vestibular function test results
* must be able to complete DVA test

Exclusion Criteria:

* Patients with central lesions will be omitted from the study because vestibular adaptation or other compensatory mechanisms may be compromised and
* Patients with visual acuity when the head is stationary of 20/60 or worse.
* Patients on medication that suppress or facilitate vestibular function will not be excluded from the study but data will be analyzed to assess the effect of medication.
* Patient who do not understand the purpose of the study and what it involves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2000-08; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Herdman, PhD, Principal Investigator — Emory University
Locations (1):
- Center for Rehabilitation Medicine, Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Herdman SJ, Tusa RJ, Blatt P, Suzuki A, Venuto PJ, Roberts D. Computerized dynamic visual acuity test in the assessment of vestibular deficits. Am J Otol. 1998 Nov;19(6):790-6. PMID 9831156
- [Result] Herdman SJ, Schubert MC, Tusa RJ. Role of central preprogramming in dynamic visual acuity with vestibular loss. Arch Otolaryngol Head Neck Surg. 2001 Oct;127(10):1205-10. doi: 10.1001/archotol.127.10.1205. PMID 11587600
- [Result] Schubert MC, Herdman SJ, Tusa RJ. Functional measure of gaze stability in patients with vestibular hypofunction. Ann N Y Acad Sci. 2001 Oct;942:490-1. doi: 10.1111/j.1749-6632.2001.tb03777.x. No abstract available. PMID 11710496
- [Result] Schubert MC, Herdman SJ, Tusa RJ. Vertical dynamic visual acuity in normal subjects and patients with vestibular hypofunction. Otol Neurotol. 2002 May;23(3):372-7. doi: 10.1097/00129492-200205000-00025. PMID 11981398
- [Result] Herdman SJ, Schubert MC, Das VE, Tusa RJ. Recovery of dynamic visual acuity in unilateral vestibular hypofunction. Arch Otolaryngol Head Neck Surg. 2003 Aug;129(8):819-24. doi: 10.1001/archotol.129.8.819. PMID 12925338
- [Result] Schubert MC, Das V, Tusa RJ, Herdman SJ. Cervico-ocular reflex in normal subjects and patients with unilateral vestibular hypofunction. Otol Neurotol. 2004 Jan;25(1):65-71. doi: 10.1097/00129492-200401000-00013. PMID 14724495
- [Result] Hall CD, Schubert MC, Herdman SJ. Prediction of fall risk reduction as measured by dynamic gait index in individuals with unilateral vestibular hypofunction. Otol Neurotol. 2004 Sep;25(5):746-51. doi: 10.1097/00129492-200409000-00017. PMID 15354006
- [Derived] Saleh M, Boukhdoud M, Boukhdoud H, Al Zein M, Salameh P. Landscape of Guillain-Barre Syndrome Interventional Clinical Trials. J Clin Neuromuscul Dis. 2023 Mar 1;24(3):119-129. doi: 10.1097/CND.0000000000000441. PMID 36809199
- [Derived] Herdman SJ, Hall CD, Schubert MC, Das VE, Tusa RJ. Recovery of dynamic visual acuity in bilateral vestibular hypofunction. Arch Otolaryngol Head Neck Surg. 2007 Apr;133(4):383-9. doi: 10.1001/archotol.133.4.383. PMID 17438254

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercises for Gaze Stabilization | Control Exercises
Started | 13 | 10
Completed | 13 | 8
Not Completed | 0 | 2
Not completed — Ten participants were entered into the c | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Exercises for Gaze Stabilization: Experimental group performed gaze stabilization exercises: adaptation and substitution exercises encorporating retinal slip and head movements
- Total: Total of all reporting groups
Arm/Group | Exercises for Gaze Stabilization | Control Exercises | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (16.5) | 64.9 (16.2) | 65.1 (16.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 7 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23
Visual acuity during head movements [Mean (Standard Deviation); unit: LogMAR] | .372 (.155) | .323 (.117) | .348 (.136)

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Acuity During Head Movement From Baseline to Discharge
Description: visual acuity is measured using a computerized system first with the head stationary and then with the head moving in yaw plane. Head velocity is measured using a rate sensor and optotype is displayed only when head velocity is between 120 and 180 degrees per second.
  The change in visual acuity was calculated from subtracting the discharge measurement from the baseline measurement (pre-intervention).
Time Frame: pre-intervention and at discharge
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Exercises for Gaze Stabilization | Control Exercises
Number analyzed (Participants) | 13 | 8
LogMAR | 0.198 (0.101) | .296 (.122)

2. Primary Outcome: Subjective Complaints: (All Pre- and Post-intervention):
Description: questionnaire
Time Frame: pre-intervention, 2 weeks, 4 weeks and at discharge
Reporting Status: Not Posted

3. Secondary Outcome: Disability Scale
Description: questionnaire
Time Frame: pre-intervention, 2 weeks, 4 weeks and at discharge
Reporting Status: Not Posted

4. Secondary Outcome: Activities Specific Balance Confidence Scale
Description: questionnaire
Time Frame: pre-intervention, 2 weeks, 4 weeks and at discharge
Reporting Status: Not Posted

5. Secondary Outcome: Symptoms Intensity for Dizziness, Oscillopsia, Disequilibrium
Description: visual analoque scales
Time Frame: pre-intervention, 2 weeks, 4 weeks and at discharge
Reporting Status: Not Posted

6. Secondary Outcome: Balance and Gait
Description: gait speed
Time Frame: pre-intervention, 2 weeks, 4 weeks and at discharge
Reporting Status: Not Posted

7. Secondary Outcome: Fall Risk (Dynamic Gait Index)
Description: performance test
Time Frame: pre-intervention, 2 weeks, 4 weeks and at discharge
Reporting Status: Not Posted

8. Secondary Outcome: Eye Movements: Scleral Search Coil
Description: eye movements are measured by having the participant sit within an electromagnetic field while wearing a scleral coil (like a contact lens but only in contact with the sclea, not the cornea); te coil moves with eye movement and distorts the electrimagnetic field
Time Frame: pre- and post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Exercises for Gaze Stabilization | Control Exercises
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercises for Gaze Stabilization (N=13) | Control Exercises (N=8)
falls (Nervous system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No